CLINICAL TRIAL: NCT05786170
Title: Early Recurrent Ischemic Lesions (ERILs) and Silent Neurologic Ischemic Lesions (SNILs) in Diffusion-weighted Magnetic Resonance Imaging (DW-MRI) - a Pilot- Observational Study Under Standard of Care (SOC)
Brief Title: ERILs Und SNILs Unter SOC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of research funding
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Christa Firbas MD, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ERILs und SNILs unter SOC
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- magnetic resonance imaging (Experimental): DW-MRI after ischemic stroke
  Interventions: Diagnostic Test: diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: diffusion-weighted magnetic resonance imaging — diffusion-weighted magnetic resonance imaging

SUMMARY:
1. How many ERILs occur in caucasian patients with LAA stroke during 7 days on standard treatment?
2. How many SNILs occur between 7 and 30 days after acute ischemic event on standard treatment?
3. How many of during acute event diagnosed lesions (ERILs) are (still) detectable after 30 days?
4. Are there relevant risk faktors for the occurence of ERILs and SNILs (eg Diabetes or Biomarkers)?

DETAILED DESCRIPTION:
In this trial, patients will be observed if they develop early recurrent ischemic lesions (= ERILs) or silent neurologic ischemic lesions (= SNILs) after acute stroke or transitoric ischemic attack (TIA) based on atherothrombosis (LAA-stroke) on standard therapy during 30 days (day 7 and day 30 after acute event) via DW-MRI (diffusion-weighted magnetic resonance imaging).

We want to investigate if diffusion-weighted imaging of silent brain infarcts occuring during standard therapy is a suitable surrogate outcome measure for interventional studies

ELIGIBILITY:
Inclusion Criteria:

* LAA stroke or TIA
* ERILs or SNILs detected in initialDW-MRI
* signed informed consent

Exclusion Criteria:

* planned surgical intervention
* iv Thrombolysis
* atrial fibrillation
* contra indications against DW-MRI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
1. How many ERILs occur in caucasian patients with LAA stroke during 7 days on standard treatment? | 7 days after acute stroke
  DW-MRI to detect lesions

SECONDARY OUTCOMES:
2. How many SNILs occur between 7 and 30 days after acute ischemic event on standard treatment and how many of during acute event diagnosed lesions (ERILs) are (still) detectable after 30 days? | 30 days after acute stroke
  DW-MRI to detect lesions